CLINICAL TRIAL: NCT00140270
Title: Evaluating the Effectiveness of a Neuromuscular and Proprioceptive Training Program to Reduce Ligamentous Knee Injuries Among Female Collegiate Soccer Players.
Brief Title: RCT of PEP Program to Reduce ACL Injuries in Female Collegiate Soccer Players
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCIPC-3185
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2005-09-01 (Estimated); Status verified 2005-08

CONDITIONS: Anterior Cruciate Ligament Rupture
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

INTERVENTIONS:
Behavioral: PEP program

SUMMARY:
This research study involves implementing and evaluating a physical training program specifically designed to reduce the risk of ligamentous knee injuries in female soccer players by incorporating proven neuromuscular and proprioceptive training concepts into a concise, on-field warm-up activity. All 283 Division I NCAA women's soccer teams were asked to participate in this research study. Those that agreed were randomized to control (usual training program) and intervention (alternative warm-up program). Both groups of teams provided investigators with participation and knee injury information during the 15 week 2002 fall soccer season. Requested information included only that which would be readily available to the certified athletic trainers (ATC) in their normal course of duties. The knee injury rates among intervention team athletes were compared with control team athletes to determine program effectiveness. Data collection is complete and the report should be submitted shortly for publication.

DETAILED DESCRIPTION:
This research study involves implementing and evaluating a physical training program specifically designed to reduce the risk of ligamentous knee injuries in female soccer players by incorporating proven neuromuscular and proprioceptive training concepts into a concise, on-field warm-up activity. All 283 Division I NCAA women's soccer teams were asked to participate in this research study. Those that agreed were randomized to control (usual training program) and intervention (alternative warm-up program). Both groups of teams provided investigators with participation and knee injury information during the 15 week 2002 fall soccer season. Requested information included only that which would be readily available to the certified athletic trainers (ATC) in their normal course of duties. The knee injury rates among intervention team athletes were compared with control team athletes to determine program effectiveness. Data collection is complete and the report should be submitted shortly for publication.

ELIGIBILITY:
Inclusion Criteria:

* Female soccer athlete on participating Division I women's soccer team

Exclusion Criteria:

* none

Min Age: 0 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4000
Dates: Start 2002-08; Study Completion 2002-12

PRIMARY OUTCOMES:
Ligamentous knee and ankle injuries;
specific interest is the ACL

CONTACTS AND LOCATIONS:
Overall Officials: Julie Gilchrist, MD, Principal Investigator — Centers for Disease Control and Prevention

REFERENCES:
- See also: site has description of the intervention under study — http://www.aclprevent.com/